CLINICAL TRIAL: NCT06876194
Title: The Effectiveness of Music on The Procedural Sedation and Analgesia Quality Among Children in The Emergency Department.
Brief Title: The Effect of Music on the Sedation Quality Among Children in the Emergency Department.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Tehran University of Medical Sciences (Other)
Responsible Party: Principal Investigator, Hadi Mirfazaelian, Associate Professor, Tehran University of Medical Sciences
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 9811307001
Record Dates: First submitted 2025-03-08; First posted 2025-03-14 (Actual); Last update posted 2025-12-08 (Actual); Status verified 2025-12

CONDITIONS: Sedation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Music (Active Comparator): A previously defined list of songs will be administered to these patients during the procedure.
  Interventions: Other: Music intervention
- No music (No Intervention)

INTERVENTIONS:
Other: Music intervention — A previously defined list of songs will be administered to these patients during the procedure.
  Arms: Music

SUMMARY:
Children presenting to the emergency department frequently experience anxiety and may undergo various painful procedures. While sedative agents are administered to these patients, they do not consistently provide adequate relief to keep the child calm and cooperative during the procedures. Implementing non-pharmacological interventions, such as music, might enhance the efficacy of sedation, resulting in a better experience for these patients and more favorable outcomes.

DETAILED DESCRIPTION:
This is an interventional single-blinded randomized clinical trial on children presenting to the emergency department of Imam Khomeini Hospital in Tehran. The estimated sample size is 42 patients in each group considering a 5% margin of error and 80% power. The efficacy of analgesia and sedation and adverse effects are measured using a predefined form. for the description of qualitative data, frequency will be used and for quantitative data, the T-Test, ANOVA, mean and SD will be employed. For examining differences between the two groups, Chi-Square, T-Test, and ANOVA will be utilized.

ELIGIBILITY:
Inclusion Criteria:

* Children between 0-14 years of age
* Requiring analgesia or sedation for medical procedures

Exclusion Criteria:

* Lack of consent from parents or legal guardian of the child
* Hearing impairment
* Any developmental disorder

Ages: 0 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 88 (Actual)
Dates: Start 2025-03-31 (Actual); Primary Completion 2025-06-08 (Actual); Study Completion 2025-07-29 (Actual)

PRIMARY OUTCOMES:
Sedation depth | Interval between start to the end of the procedure, an average of 30 minute
  Using the Pediatric Sedation State Scale (PSSS), we will assess the sedation depth of the children.

SECONDARY OUTCOMES:
Adverse effect | Interval between injection to the end of recovery for 2 hours
  Using standard definitions, the adverse effects will be assessed.
Recovery condition | Interval between the end of the procedure to the full recovery for 2 hours
  using a three-level scale, we will assess the child recovery condition.
Physicians' satisfaction | Interval between start to the end of the procedure, an average of 30 minute
  We will use the 5-level Likert scale to assess the physicians' satisfaction with the sedation and procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Hadi Mirfazaelian, MD, Principal Investigator — Tehran University of Medical Sciences
Locations (1):
- IKHC, Tehran, Iran

IPD SHARING:
Plan to Share IPD: No
The information is not allowed to be shared.